CLINICAL TRIAL: NCT04900714
Title: Minimizing Lung Injury During Laparoscopy in Steep Trendelenburg Position
Acronym: optiPEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20/40/516; 1378 (Other: EDGE); 20/40/516 (Other: IRB)
Record Dates: First submitted 2020-09-24; First posted 2021-05-25 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Atelectasis
Keywords: Positive-Pressure Respiration; Respiratory Mechanics; positive end-expiratory pressure
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Blood Gas Analysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decremental PEEP (Experimental): Every participant will be exposed to a stepwise decremental PEEP.
  Interventions: Procedure: Decremental PEEP; Diagnostic Test: Lung ultrasound score; Diagnostic Test: Blood gas analysis; Diagnostic Test: Registration of respiratory mechanics; Diagnostic Test: Evaluation of dead space

INTERVENTIONS:
Procedure: Decremental PEEP — High PEEP to low PEEP.
Diagnostic Test: Lung ultrasound score — lung ultrasound to determine the extend of atelectasis. Uses validated lung ultrasound score.
Diagnostic Test: Blood gas analysis — Blood gas analysis to determine arterial oxygen tension
Diagnostic Test: Registration of respiratory mechanics — Pressures and volumes will be registered by the Fluxmed respiratory monitor (MBMED, Argentina)
Diagnostic Test: Evaluation of dead space — Dead space will be measured non-invasively using volumetric capnography on the FluxMed respiratory monitor (MBMED, Argentina)

SUMMARY:
The investigators hypothesize that the level of PEEP is often suboptimally applied in certain operative conditions, such as in laparoscopy with head down (Trendelenburg) positioning. This can result in excessive levels of lung stress and postoperative pulmonary complications.

In patients with steep Trendelenburg and a pneumoperitoneum, the investigators aim to

1. measure apical versus basal atelectasis using the lung ultrasound score
2. compare lung ultrasound scores at different PEEP levels
3. compare respiratory mechanics at the different PEEP levels
4. contrast the optimal PEEP level to standard practice
5. provide guidance to optimal PEEP titration in this setting for the clinician

DETAILED DESCRIPTION:
The investigators hypothesize that the level of positive end-expiratory pressure (PEEP) is often incorrectly applied in certain operative conditions, such as in laparoscopy with head down (Trendelenburg) positioning. This can result in excessive levels of lung stress and postoperative pulmonary complications.

Incorrect intra-operative ventilator management can be harmful for the patient, potentially leading to postoperative pulmonary complications and ventilator-induced lung injury. During routine anesthesia procedures, most anesthetists will set the ventilator by rule of thumb with a PEEP of 4-6 cmH2O, a tidal volume of 6-8 ml/kg of ideal body weight and a frequency of 10-15 breaths per minute in order to provide lung protective ventilation. However, due to recent advances in surgical practice, patients are more frequently placed in non- physiological states, such as Trendelenburg position up to 30° with concurrent pneumoperitoneum and intra-abdominal pressures of 15mmHg or higher, as in for example robot-assisted radical prostatectomy or gynecological procedures. This extreme positioning and increased intra-abdominal pressure can have a significant effect on respiratory mechanics and can potentially result in excessive lung stress. The changes in applied positive pressure ventilation will result in changes of regional ventilation: both an increased amount of atelectasis and an increased amount of regional hyperinflation are observed in this setting. The ideal PEEP level balances the recruitment of atelectasis versus excessive hyperinflation. These changes in regional ventilation can be assessed by lung ultrasound. The lung ultrasound score can distinguish atelectasis from normal aeration in the different lung regions of interest.

This project is designed as a single center cohort study. Non-obese (BMI < 30kg/m2), lung-healthy non-pregnant, non-smoking individuals without right sided heart failure, scheduled for elective laparoscopy of the lower abdomen, will be recruited. Standardized induction and maintenance with propofol TCI (3-6μg/l plasma concentration as calculated by the Marsh model), sufentanil (0.2μg/kg) and rocuronium (0.6mg/kg) will be provided. Neuromuscular blockade will be monitored using a train-of-four (TOF) monitor and kept with a TOF count < 1 throughout the study using additional doses if indicated. A radial arterial line will be placed. Mechanical ventilation will be provided in volume control mode with a tidal volume of 4-6 ml/kg of ideal body weight (IBW) aiming for a driving pressure ≤ 15cmH2O, a starting PEEP of 5cmH2O, a frequency of 12-18 breaths per minute titrated to the end-tidal CO2 measurement and an initial FiO2 of 0.4. An esophageal balloon catheter with pressure sensor will be used to calculate transpulmonary pressures. The balloon and pressure sensor will be calibrated as per manufacturers guideline. Respiratory parameters will be recorded and saved for later evaluation using the FluxMed GrT monitor and software (MBMED, Argentina). After inflation of the pneumoperitoneum, lung ultrasound will be performed bilaterally at the midclavicular line between the second and third ribs, at the posterior axillary line above the level of T4 and at the posterior axillary line closely superior to the diaphragm, thus retaining 6 ultrasound loops which will be saved for post-hoc lung ultrasound scoring. The lung ultrasound measurements will be repeated at different decremental levels of PEEP: 15, 10, 5 and 0 cmH2O respectively. Arterial blood gas analysis will be performed before insufflation of the pneumoperitoneum and repeated at each level of PEEP. A minimum of 4 minutes equilibration time will be provided after changing PEEP.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopy in the Trendelenburg (head-down) position

Exclusion Criteria:

* smoker
* lung disease (e.g. asthma, COPD, emphysema)
* BMI > 30 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Lung ultrasound score | Perioperatively
  Lung ultrasound score per level of PEEP (15-10-5-0 cmH2O). The score is dimensionless. A cumulative count is calculated for each level of PEEP by adding the scores from the 6 scanned lung regions together.
  The lung ultrasound score is a measure of atelectasis.

SECONDARY OUTCOMES:
Transpulmonary pressure (cmH2O) | Perioperatively
  Transpulmonary pressure per level of PEEP (15-10-5-0 cmH2O). Transpulmonary pressure is calculated as plateau airway pressure minus esophageal pressure (at the same timepoint).
  Plateau airway pressures (cmH2O) are measured at the ventilator during an inspiratory pause.
  Esophageal pressures (cmH2O) are measured with an esophageal balloon and pressure transducer.
  Esophageal pressures are proven to correlate closely to pleural pressures. The Fluxmed device (MBMED, Argentina) is used to capture pressures and volumes at the ventilator.
Driving pressure (cmH2O) | Perioperatively
  Driving pressures per level of PEEP (15-10-5-0 cmH2O). Driving pressure (cmH2O) is calculated as plateau airway pressure minus positive end-expiratory pressure (PEEP).
  Plateau airway pressures (cmH2O) are measured at the ventilator during an inspiratory pause.
  PEEP (cmH2O) is measured at the ventilator at end-expiration. The Fluxmed device (MBMED, Argentina) is used to capture pressures and volumes at the ventilator.
Dynamic pulmonary compliance (ml/cmH2O) | Perioperatively
  Dynamic pulmonary compliance per level of PEEP (15-10-5-0 cmH2O). The dynamic pulmonary compliance is calculated as tidal volume divided by the driving pressure.
  Tidal volumes (ml) are measured at the ventilator. Driving pressures are calculated as mentioned in the description of outcome 3. The Fluxmed device (MBMED, Argentina) is used to capture pressures and volumes at the ventilator.
P/F ratio (Horowitz index, mmHg / %) | Perioperatively
  Ratio of the arterial oxygen tension (mmHg) divided by the fraction of inspired oxygen (%) per level of PEEP (15-10-5-0 cmH2O).
  The arterial oxygen tension is measured at a point-of-care blood gas analyzer (Roche Cobas, Basel, Swiss) The inspiratory oxygen fraction (%) is measured at the ventilator.
Dead space | Perioperatively
  Median dead space per level of PEEP (15-10-5-0 cmH2O).

CONTACTS AND LOCATIONS:
Overall Officials: Vera Saldien, MD, PhD, Principal Investigator — Head of the department of anesthesiology; Tom Schepens, MD, PhD, Study Chair — Anesthetist/intensivist; Gregory De Meyer, MD, Study Chair — Anesthetist in training; Stuart G Morrison, MD, Study Director — Staff anesthetist
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Meyer GRA, Morrison SG, Saldien V, Jorens PG, Schepens T. Minimizing Lung Injury During Laparoscopy in Head-Down Tilt: A Physiological Cohort Study. Anesth Analg. 2023 Oct 1;137(4):841-849. doi: 10.1213/ANE.0000000000006325. Epub 2022 Dec 14. PMID 36729514